CLINICAL TRIAL: NCT05179616
Title: Pforzheim Tricuspid Valve Registry: A Real-world Observational Trial Evaluating Outcomes in Patients Treated With the Abbott TriClip™ Device in Helios Klinikum Pforzheim
Brief Title: Pforzheim Tricuspid Valve Registry - Outcomes of Percutaneous Tricuspid Valve Repair
Status: Recruiting | Type: Observational
Sponsor: Helios Klinikum Pforzheim (Other)
Responsible Party: Principal Investigator, Patrascu Alexandru, Principal Investigator, Helios Klinikum Pforzheim
Other Study IDs: PF-TriValve
Record Dates: First submitted 2021-11-27; First posted 2022-01-05 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Tricuspid Regurgitation; Right Heart Failure; Cardiac Remodeling, Ventricular; Cardiac Remodeling, Atrial
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure; Ventricular Remodeling; Atrial Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Patients suffering from symptoms of right heart failure due to high-grade tricuspid regurgitation
  Interventions: Procedure: Transcatheter edge-to-edge tricuspid valve repair

INTERVENTIONS:
Procedure: Transcatheter edge-to-edge tricuspid valve repair — Percutaneous edge to edge repair of tricuspid valve using the TriClip system

SUMMARY:
The Pforzheim Tricuspid Valve Registry study is designed to confirm the safety and performance of the TriClip™ device in a contemporary real-world setting in critically ill patients. The observational trial is a prospective, single arm, open-label, single-center, post market registry.

DETAILED DESCRIPTION:
Significant tricuspid regurgitation is a common finding in elderly patients, with an incidence of 5.6% after the age of 70 years, according to the Framingham Heart Study. TR is an independent predictor for adverse prognosis and has limited treatment options. Tricuspid valve (TV) intervention is indicated when symptomatic TR-related right heart failure (RHF) is present. However, the surgical risk is usually deemed to be too high due to the presence of advanced age, pulmonary hypertension, right ventricular (RV) impairment, major organ failure and other co-morbidities. Moreover, isolated tricuspid valve surgery has an in-hospital mortality of approx. 8,7%, according to recent data.

High TR prevalence, coupled with low incidence of isolated TV surgery, has created a considerable population in need of alternative, percutaneous therapies to improve outcomes. Recently, a variety of interventional procedures and devices have been developed which simulate different surgical approaches like suture or ring annuloplasty, coaptation enhancement, neochordae repair, or even valve replacement. Among them, coaptation devices attempt to correct leaflet malcoaptation by using the edge-to-edge clip technique, similar to treatment of functional mitral regurgitation. To date, most TTVR interventions have been performed off-label with the MitraClip device.

Last year, the first TR dedicated device (TriClipTM, Abbott Medical) has been approved (CE mark), after showing good feasibility, safety and effectiveness, and meanwhile sustained and marked clinical benefit with low mortality after 12 months.

Although most TTVR studies have enrolled high-risk cohorts, criteria for patient selection and timing of intervention have yet to be defined. Based on scientific surgical data, it seems reasonable to expect poorer outcomes in patients with several comorbidities, advanced cardiac remodeling and RHF-related major organ dysfunction e.g., renal and hepatic function impairment. Whether or not this assumption can be extrapolated to TTVR needs to be investigated.

In this registry, the investigators aim to evaluate if percutaneous therapy with the TriClip system is safe and effective in patients at high and prohibitive risk and wether or not procedural success is the main determinant of short-, mid- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (>=18 years age) have severe tricuspid regurgitation and are symptomatic despite medical therapy.
* Subjects eligible to receive the TriClip™
* Subjects must provide written informed consent prior to study procedure.

Exclusion Criteria:

* Subjects participating in another clinical study that may impact the follow-up or results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have symptomatic severe tricuspid regurgitation despite medical therapy and are eligible to receive the TriClip™
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | at 12 months
  One-grade reduction of tricuspid regurgitation

SECONDARY OUTCOMES:
Change in quality of life | at 12 months
  NYHA class
Change in functional capacity | at 12 months
  6-minute walk test
Major organ system functional change | at12 months
  Renal and hepatic function as assessed by following lab values: creatinine, glomerular filtration rate, aspartate transaminase, alanine aminotransferase and bilirubine

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Ott, MD, PhD, Principal Investigator — Helios Klinikum Pforzheim
Locations (1):
- Helios Klinikum Pforzheim, Pforzheim, Germany

IPD SHARING:
Plan to Share IPD: No